CLINICAL TRIAL: NCT02512510
Title: A Phase 3, 12-week, Randomized, Double-blind Placebo-controlled Parallel Group Study of Nebulized TD-4208 in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy Study of Nebulized TD-4208 for Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0127
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TD-4208-1 (Active Comparator): 88 mcg
  Interventions: Drug: TD-4208
- TD-4208-2 (Active Comparator): 175 mcg
  Interventions: Drug: TD-4208
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-4208
  Other Names: revefenacin
  Arms: TD-4208-1; TD-4208-2
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the effectiveness and safety of TD 4208, an investigational drug being developed to treat people with moderate to very severe COPD, compared to placebo, a treatment without activity.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female subject 40 years of age or older

Exclusion Criteria:

* Females who are pregnant, lactating, breast-feeding or planning to become pregnant during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Palmetto Medical Research Associates L.L.C., Easley, South Carolina, United States

REFERENCES:
- [Derived] Donohue JF, Ferguson GT, Ohar JA, Lombardi DA, Schneider RF, Johnson K. Improvements in health status with revefenacin, a once-daily, nebulized, long-acting muscarinic antagonist for chronic obstructive pulmonary disease. Respir Med. 2023 Mar;208:107123. doi: 10.1016/j.rmed.2023.107123. Epub 2023 Jan 18. PMID 36681255
- [Derived] Lo A, Borin MT, Bourdet DL. Population Pharmacokinetics of Revefenacin in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2021 Mar;60(3):391-401. doi: 10.1007/s40262-020-00938-3. PMID 33124005
- [Derived] Donohue JF, Kerwin E, Barnes CN, Moran EJ, Haumann B, Crater GD. Efficacy of revefenacin, a long-acting muscarinic antagonist for nebulized therapy, in patients with markers of more severe COPD: a post hoc subgroup analysis. BMC Pulm Med. 2020 May 11;20(1):134. doi: 10.1186/s12890-020-1156-4. PMID 32393215

RESULTS

PARTICIPANT FLOW:
Groups:
- TD-4208-1: 88 mcg
  TD-4208
- TD-4208-2: 175 mcg
  TD-4208
Period: Overall Study
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
Started | 205 | 197 | 209
Completed | 163 | 162 | 157
Not Completed | 42 | 35 | 52

BASELINE CHARACTERISTICS:
Population: 611 subjects randomized. 1 subject was not dosed and was thus not included in any analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo | Total
Number analyzed (Participants) | 205 | 197 | 208 | 610
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 121 | 106 | 115 | 342
  >=65 years | 84 | 91 | 93 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.81) | 63.6 (9.19) | 63.5 (8.91) | 63.4 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 95 | 111 | 308
  Male | 103 | 102 | 97 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 12 | 39
  Not Hispanic or Latino | 188 | 186 | 194 | 568
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 21 | 20 | 58
  White | 186 | 171 | 188 | 545
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 205 | 197 | 208 | 610
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 97 | 94 | 95 | 286
  Former Smoker | 108 | 103 | 113 | 324

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 on Day 85
Time Frame: Baseline and Day 85
Population: Intent-to-treat (ITT) analysis set
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
Number analyzed (Participants) | 152 | 154 | 150
mL | 115.58 (18.637) | 102.90 (18.542) | -44.92 (18.841)

2. Secondary Outcome: Summary of Trough FEV1 Overall Treatment Effect From Day 15 to Day 85
Time Frame: Days 15 to 85
Measure: Mean (Standard Error); unit: mL
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
Number analyzed (Participants) | 189 | 181 | 187
mL | 83.9 (3.14) | 87.1 (3.21) | -39.9 (3.15)

3. Secondary Outcome: Summary of Change From Baseline to Peak FEV1 After First Dose
Time Frame: 0-2 hours after First Dose Day 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
Number analyzed (Participants) | 204 | 196 | 208
mL | 218.65 (10.291) | 216.84 (10.248) | 88.22 (10.092)

4. Secondary Outcome: Summary of Rescue Medication Use: Puffs Per Day
Time Frame: 1-3 Months
Measure: Least Squares Mean (Standard Error); unit: Puffs per Day
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
Number analyzed (Participants) | 202 | 196 | 203
Puffs per Day | 2.00 (0.207) | 2.38 (0.204) | 2.54 (0.206)

5. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Proportion of Responders on Day 85
Description: A Responder is defined as someone who experienced a decrease in SGRQ score of 4 or more units
Time Frame: Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
Number analyzed (Participants) | 145 | 149 | 140
Participants | 67 | 67 | 54

6. Secondary Outcome: Percentage of Albuterol Rescue-free 24-hour Periods
Time Frame: 1-3 Months
Measure: Least Squares Mean (Standard Error); unit: Percentage of 24hr periods
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
Number analyzed (Participants) | 205 | 197 | 207
Percentage of 24hr periods | 44.79 (2.800) | 43.26 (2.769) | 37.23 (2.766)

ADVERSE EVENTS:
Time Frame: From signing of ICF through the final follow-up assessment, Day 85.
Arm/Group | TD-4208-1 | TD-4208-2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/205 | 1/197 | 0/209
Serious Adverse Events (participants affected / at risk) | 11/205 | 5/197 | 7/209
Other Adverse Events (participants affected / at risk) | 59/205 | 62/197 | 52/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TD-4208-1 (N=205) | TD-4208-2 (N=197) | Placebo (N=209)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrolvascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Victim of homicide (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TD-4208-1 (N=205) | TD-4208-2 (N=197) | Placebo (N=209)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 21 (21) | 25 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 10 (10) | 9 (9)
Headache (Nervous system disorders) | 14 (14) | 8 (8) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 10 (10) | 5 (5)
Nasopharyngitis (Infections and infestations) | 7 (7) | 9 (9) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.